CLINICAL TRIAL: NCT05323695
Title: Implementation of a Depression Screening Intervention at a Transgender Health Clinic in Thailand
Acronym: CHIMERA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Thai Red Cross AIDS Research Centre (Other)
Collaborators: amfAR, The Foundation for AIDS Research (Other); National Institutes of Health (NIH) (NIH); Fogarty International Center of the National Institute of Health (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: IHRI008; D43TW011302 (NIH)
Record Dates: First submitted 2021-07-08; First posted 2022-04-12 (Actual); Last update posted 2024-11-26 (Actual); Status verified 2024-11

CONDITIONS: Depressive Symptoms
Keywords: Depression; Transgender women
MeSH Terms: conditions — Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Depression Screening Intervention (Other): All eligible participants will be screened using the Patient Health Questionnaire-2 (PHQ-2) for depression. If screened positive, participants will be further screened with Patient Health Questionnaire-9 (PHQ-9).
  Interventions: Behavioral: Depression Screening Intervention

INTERVENTIONS:
Behavioral: Depression Screening Intervention — All participants will be screened for depression using PHQ-2 and PHQ-9. Those screened positive for PHQ-2 but decline further screening with PHQ-9 will be assisted for further assessment or care. Those with mild to severe symptoms (score of 7 or higher on PHQ-9) will be assisted for further assessment or care with a psychiatrist.

SUMMARY:
The study aims to develop and implement a depression screening intervention into routine HIV and sexual health service provision at a transgender health clinic in Thailand, and to explore the facilitators, barriers, feasibility and acceptability of the screening implementation.

DETAILED DESCRIPTION:
The study will follow a mixed-methods approach that will incorporate quantitative and qualitative components. Aim 1 will involve the development and implementation of depression screening intervention at Tangerine Clinic. Aim 2 will involve semi-structured interviews with a purposive subset of participants who received the intervention and healthcare providers to explore the multilevel facilitators, barriers, feasibility and acceptability of the screening implementation. Aim 3 will evaluate the proportion of participants who are offered, accept, and receive the peer-led depression screening intervention, and the proportion who screen positive.

ELIGIBILITY:
Inclusion Criteria:

1. Thai nationality
2. Transgender women ≥18 years
3. Attending the Tangerine Clinic for routine care visits during the intervention period.
4. Can be a new or returning clients.

Exclusion Criteria:

1. Transgender women currently receiving care for a mental health diagnosis will be excluded from participating in this study.

Inclusion Criteria for healthcare providers:

1. Currently working at the Tangerine Clinic
2. Can be medical doctors, nurses, peer counselors and other members of the clinic management team involved in the routine delivery of HIV and health services to Transgender women.

Exclusion criteria for healthcare providers

1. Not willing to participate in this study

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 317 (Actual)
Dates: Start 2021-10-11 (Actual); Primary Completion 2023-02-15 (Actual); Study Completion 2024-07-02 (Actual)

PRIMARY OUTCOMES:
Intervention Acceptability: Number of participants who accepted intervention | Day 1
  Acceptability will be measured by the number of clients who were offered and accepted the intervention.
Intervention Acceptability: Participants' perspective of the intervention through in-depth interviews | Day 1
  Acceptability will be assessed qualitatively through post-intervention in-depth interviews.
Intervention Acceptability: Participants' perspective of the intervention through focus group discussion | Day 1
  Acceptability will be assessed qualitatively through post-intervention focus group discussion.
Intervention Feasibility: Number of intervention completed | Day 1
  Feasibility will be measured by number of intervention completed. Point estimates of >50% of participants completed is considered as the minimum criteria for feasibility.
Intervention Feasibility: Participants' perspective of the intervention through in-depth interviews | Day 1
  Feasibility will be assessed qualitatively through post-intervention in-depth interviews.
Intervention Feasibility: Participants' perspective of the intervention through focus group discussion. | Day 1
  Feasibility will be assessed qualitatively through post-intervention focus group discussion.
Number of participants screening positive for depression | Day 1
  Screening positive is defined as scoring 7 or greater on PHQ-9. The total possible score for PHQ-9 is 27, with 0-6 being minimum and indicating no depressive symptoms, 7-12 mild depression, 13-18 moderate depression, and 19-27 severe depression.

CONTACTS AND LOCATIONS:
Overall Officials: Rena Janamnuaysook, Principal Investigator — Institute of HIV Research and Innovation
Locations (1):
- Institute of HIV Research and Innovation, Pathum Wan, Bangkok, Thailand

REFERENCES:
- [Background] Anand T, Nitpolprasert C, Kerr SJ, Muessig KE, Promthong S, Chomchey N, Hightow-Weidman LB, Chaiyahong P, Phanuphak P, Ananworanich J, Phanuphak N. A qualitative study of Thai HIV-positive young men who have sex with men and transgender women demonstrates the need for eHealth interventions to optimize the HIV care continuum. AIDS Care. 2017 Jul;29(7):870-875. doi: 10.1080/09540121.2017.1286288. Epub 2017 Feb 3. PMID 28158952
- [Background] Schulman JK, Erickson-Schroth L. Mental Health in Sexual Minority and Transgender Women. Med Clin North Am. 2019 Jul;103(4):723-733. doi: 10.1016/j.mcna.2019.02.005. PMID 31078203
- [Background] Kroenke K, Spitzer RL, Williams JB. The Patient Health Questionnaire-2: validity of a two-item depression screener. Med Care. 2003 Nov;41(11):1284-92. doi: 10.1097/01.MLR.0000093487.78664.3C. PMID 14583691
- [Background] Poteat T, Scheim A, Xavier J, Reisner S, Baral S. Global Epidemiology of HIV Infection and Related Syndemics Affecting Transgender People. J Acquir Immune Defic Syndr. 2016 Aug 15;72 Suppl 3(Suppl 3):S210-9. doi: 10.1097/QAI.0000000000001087. PMID 27429185
- [Background] Rodriguez-Munoz MF, Castelao Legazpi PC, Olivares Crespo ME, Soto Balbuena C, Izquierdo Mendez N, Ferrer Barrientos FJ, Huynh-Nhu L. [PHQ-2 as First Screening Instrument of Prenatal Depression in Primary Health Care, Spain]. Rev Esp Salud Publica. 2017 Jan 30;91:e201701010. Spanish. PMID 28134236
- [Background] Martinez P, Soto-Brandt G, Brandt S, Guajardo V, Rojas G. [Validation of patient health Questionnaire-2 to detect depressive symptoms in diabetic or hypertensive patients]. Rev Med Chil. 2020 Nov;148(11):1614-1618. doi: 10.4067/S0034-98872020001101614. Spanish. PMID 33844767
- [Background] Baral S, Logie CH, Grosso A, Wirtz AL, Beyrer C. Modified social ecological model: a tool to guide the assessment of the risks and risk contexts of HIV epidemics. BMC Public Health. 2013 May 17;13:482. doi: 10.1186/1471-2458-13-482. PMID 23679953